CLINICAL TRIAL: NCT06448767
Title: The Effect of a Multispecies Probiotics on Autism Symptoms in Children
Acronym: PROBAUT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Winclove Probiotics B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KB/151/2023
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Probiotics
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multispecies probiotics group (Experimental): 55 participants
  Interventions: Dietary Supplement: Multispecies probiotics
- Control group (Placebo Comparator): 55 participants
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Multispecies probiotics — Multispecies probiotics consisting of Bacillus subtilis W201, Bifidobacterium infantis W17, Bifidobacterium lactis W51, Lactobacillus acidophilus W37, Lactobacillus brevis W63, Lactobacillus rhamnosus W140, Lactococcus lactis W19, Propionibacterium freudenreichii W200 at a dose of 5x10^9 Colony Forming Units (CFU), once daily, orally.
  Arms: Multispecies probiotics group
Other: Placebo — Placebo identical in taste, smell and color to the multispecies probiotics.
  Arms: Control group

SUMMARY:
In this trial, the investigators aim to evaluate the impact of a multispecies probiotic consisting of Bacillus subtilis W201, Bifidobacterium infantis W17, Bifidobacterium lactis W51, Lactobacillus acidophilus W37, Lactobacillus brevis W63, Lactobacillus rhamnosus W140, Lactococcus lactis W19, Propionibacterium freudenreichii W200, on the severity of autism symptoms, quality of life, gastrointestinal symptoms, sleep disturbances, parental stress levels and urinary p-cresol concentrations in children with Autism Spectrum Disorder aged 7 to 15 years.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled clinical trial. One hundred and ten children aged 7 to 15 years diagnosed with Autism Spectrum Didorder will be randomly assigned in a 1:1 ratio to receive either a multispecies probiotics or a placebo for 12 weeks. The probiotic mixture contains 5 x 10^9 colony forming units per dose consisting of Bacillus subtilis W201, Bifidobacterium infantis W17, Bifidobacterium lactis W51, Lactobacillus acidophilus W37, Lactobacillus brevis W63, Lactobacillus rhamnosus W140, Lactococcus lactis W19, Propionibacterium freudenreichii W200.

The primary outcome will be the assessment of core autism symptoms using the Autism Symptom Rating Scales (ASRS). The secondary outcomes will include: the quality of life measured by the Quality of Life in Autism Part A questionnaire (QoLA-A), evaluations of sleep impairments using Children Sleep Habit Questionnaire - Abbreviated (CSHQ-A), parental stress levels using Parenting Stress Index-III (PSI-III), gastrointestinal symptoms using Gastrointestinal Symptom Rating Scale (GSRS), and urinary p-cresol levels. These outcomes will be assessed twice: at baseline and after 12 weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ASD according to the Diagnostic and Statistical Manual of Mental Disorders, the fifth edition (DSM-5) or International Classification of Diseases, Tenth Revision (ICD-10).
2. Children either not taking any medication or receiving the same medication for the last 2 months.
3. Patients, or their parents/caregivers, are willing to provide written informed consent, proceed with nutritional supplements throughout the 3-month trial, refrain from starting any kind of special diet for the duration of the study, and complete the questionnaires at two time points during the study.

Exclusion Criteria:

1. Use of antibiotics in the previous 2 months before enrolling (excluding topical antibiotics).
2. Use of probiotics or synbiotics within the previous 2 months.
3. History of intolerance or allergy to probiotics, synbiotics or any other study product component.
4. Surgery with bowel resection or short bowel syndrome.
5. Children with severe immunodeficiency.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
The Autism Spectrum Rating Scales (ASRS) | 0-3 months
  Assessment of the severity of ASD symptoms. Scores are reported as percentiles, with higher values indicating greater symptom severity.

SECONDARY OUTCOMES:
The Parenting Stress Index, 4th Edition (PSI-4) / SIPA (Stress Index for Parents of Adolescents) | 0-3 months
  Assessment of the parenting stress intensity. The level of parental stress will be assessed using the PSI-4 questionnaire if the child is under 11 years old, or the SIPA if the child is 11 years or older. Scores range from 101 to 505 points for the PSI-4 and 90 to 450 points for the SIPA. Higher scores indicate higher level of stress.
Children Sleep Habit Questionnaire - Abbreviated (CSHQ-A) | 0-3 months
  Assessment of the sleep impairments. Scores range from 0 to 154 points, with higher values indicating a greater severity of sleep disturbances.
The Quality of Life in Autism Part A (QoLA-A) | 0-3 months
  Assessment of the quality of life of parents of children with ASD. Scores range from 28 to 140 points, with higher values reflecting a better quality of life.
Gastrointestinal Symptom Rating Scale (GSRS) | 0-3 months
  Assessment of the severity of gastrointestinal symptoms. Scores range from 15 to 105 points, with higher values indicating greater severity of gastrointestinal symptoms.
P-cresol levels in urine samples | 0-3 months
  Assessment of the level of p-cresol in urine samples.

CONTACTS AND LOCATIONS:
Overall Officials: Maja Kotowska, MD, Principal Investigator — Department of Paediatrics, The Medical University of Warsaw, Poland
Locations (1):
- Department of Paediatrics, The Medical University of Warsaw, Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kotowska-Babol M, Konowalek L, Szajewska H, Lukasik J. Effect of multispecies probiotics on autism symptoms: protocol for a randomized controlled trial (PROBAUT). Trials. 2025 Dec 20;26(1):573. doi: 10.1186/s13063-025-09373-w. PMID 41422017